CLINICAL TRIAL: NCT04939974
Title: Evaluation of the Efficacy of Oral Probiotics Supplementation in Children With Autism Spectrum Disorders (ASDs): a Randomized Double Blind, Placebo Controlled Trial
Brief Title: Probiotic in Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Prof, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: probiotic autism
Record Dates: First submitted 2021-06-18; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic (Active Comparator): The probiotic preparation selected for this study will contain use three species of probiotic bacterias namely Lactobacillus rhamnosus - ATCC 21052, Lactobacillus plantarum - ATCC 8014 and Bifidobacterium longum subsp. Infantis-ATCC 15707 at the dose of one billion (10 9 ) CFU/g of product (Total 3x10 9 CFU/g).
  Interventions: Dietary Supplement: probiotic
- placebo (Placebo Comparator): Placebo packet same in colour, smell and constituent to that of placebo one packet daily for 24 weeks
  Interventions: Dietary Supplement: probiotic

INTERVENTIONS:
Dietary Supplement: probiotic — The probiotic preparation selected for this study will contain use three species of probiotic bacterias namely Lactobacillus rhamnosus - ATCC 21052, Lactobacillus plantarum - ATCC 8014 and Bifidobacterium longum subsp. Infantis-ATCC 15707 at the dose of one billion (10 9 ) CFU/g of product (Total 3x10 9 CFU/g).

SUMMARY:
One suitable probiotic packet will be administered to one group and placebo to another group of autism children and improvement in CARS will be monitored

ELIGIBILITY:
Inclusion Criteria:

1. All children diagnosed with Autistic Spectrum Disorders by DSM 5 criteria
2. Aged: 2-18 years.
3. Normal hearing (clinically or whenever required by Oto-acoustic emission / automated Brainstem evoked response audiometry)
4. Preferably patients from Delhi-NCR or ready to come for follow up -

Exclusion Criteria:

* On standard treatment and care for more than 12 weeks 2. Received in last 12 weeks or currently on any complementary and/or alternate therapy including dietary therapy 3. Associated chronic systemic illness 4. Known allergy to any component of probiotic supplement

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
change in childhood autism rating scale at 24 weeks as compared to baseline | 24 weeks
  change in childhood autism rating scale at 24 weeks as compared to baseline

IPD SHARING:
Plan to Share IPD: No